CLINICAL TRIAL: NCT01891552
Title: Observational Study on Second Line Treatment of Colorectal Liver Metastases (KRas wt) by Hepatic Intra-arterial Chemoembolization With Dc Beads 70-150 μm Microspheres Preloaded With Irinotecan 200 Mgr Plus Systemic Cetuximab
Brief Title: Observational Study on Second Line Treatment of Liver Metastases With DEBIRI and Cetuximab
Acronym: TACETUX
Status: Completed | Type: Observational
Sponsor: International Group of Endovascular Oncology (Other)
Responsible Party: Principal Investigator, Giammaria Fiorentini, Dr., International Group of Endovascular Oncology
Other Study IDs: TACETUX01
Record Dates: First submitted 2013-06-26; First posted 2013-07-03 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Colon Cancer Liver Metastasis
Keywords: Colon Cancer, Liver Metastasis, DEBIRI, cetuximab, efficacy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Tacetux: DEBIRI+ CETUXIMAB ADMINISTRATION
- DEBIRI: only DEBIRI treatment

SUMMARY:
* The recently introduced chemoembolization has been considered to be a very attractive new method in terms of response in the treatment of liver metastases from colon cancer carcinoma (LM-CRC). It appears to be particularly useful if carried out with the new embolization materials.
* An 80% response rate was reported using TACE with Irinotecan pre-loaded Beads in patients with liver metastases from colon cancer, who had been pretreated with 2 or more lines of chemotherapy.
* Since a greater activity was attained by a combination of Cetuximab and Irinotecan versus Cetuximab in monotherapy, the European Agency for the Evaluation of Medicinal Products (EMEA) has granted authorization to the use of Cetuximab in association with irinotecan in the treatment of irinotecan-refractory CRC-LM.
* In this study we want to collect data on on time to progression and tolerability using DEBIRI+Cetuximab in LM-CRC

DETAILED DESCRIPTION:
This is an observational study and the treatment is related to the experiences and economical availability of each center.

Primary objective: To collect data on time to progression (local and/or distant progression) after administration of Dc-Beads microspheres preloaded with Irinotecan 200 mgr via hepatic intra-arterial locoregional delivery (TACE) in/without association with standard weekly therapy with Cetuximab.

Secondary objectives: To collect data on tolerability of treatment and improvement of quality of life (Edmonton Symptom Assessment System (ESAS))

Treatment under observation :

Program A ( for all patients)

Day +1:

Lobar Infusion (lobe with dominant disease) of Irinotecan 100 mg preloaded into 2 ml of 70-150 µm M1 microspheres.

Second lobar infusion of Irinotecan 100 mg preloaded into 2 ml of 70-150 µm M1 microspheres can be administered at the same time contralaterally or in a further TACE.

Day +30: The above procedure is repeated. Day +90: In case of response, a third administration following the above procedures will be repeated

Program B ( for Centers in which Cetuximab is available) 5.2 Cetuximab administered as per standard scheme: Day -15: loading dose with 400 mg/mq i.v. over a 2-hour period Day +21 and subsequent weekly administrations: 250 mg/mq i.v. over a one hour period.

It is pointed out that administration of Cetuximab will be continued following the timeline of the first infusion relative to the intra-arterial administration.

Evaluation of response

Response must be assessed by repeating the following examinations at Day 30, Day 90 and Day 120 after start of treatment:

Chest-abdomen CAT scan with and without contrast medium (refer to Section 4). Evaluation will be based on the Response Evaluation Criteria In Solid Tumors (RECIST) cancer markers (CEA, Carbohydrate Antigen (CA) 19.9)

Assessment of quality of life The Edmonton Symptom Assessment System (ESAS) is used to monitor health conditions and quality of life.

The questionnaire must be filled in by the patient unaided by family members or by health care personnel, over a period of about 15 minutes. Assessment of quality of life will be performed during the baseline visit and at Day 30, Day 60 and Day 120 from start of treatment.

It is important for the questionnaire to be completed by the patient before undergoing the physical examination, in other words before discussing with the physician about any examinations which might give an indication of the favorable or unfavorable course of the disease. In providing the questionnaire to the patient, the physician will explain how to complete it without discussing the contents of the questions, and once the patient has completed the questionnaire, the physician will check that all questions have been answered.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable hepatic metastases from colorectal carcinoma (CRC-LM)
2. Progression of disease after first line therapy containing Irinotecan completed at least one month previously
3. Performance status (PS) 0-2
4. Biochemistry parameters within normal limits (ALT and gamma glutamyl transpeptidase not exceeding three times the upper limit of normal, total bilirubin not exceeding 2.5 mg/ml)
5. Adequate information and subsequent written informed consent
6. Life expectancy > 3 months
7. Patients K-RAS wild type

Exclusion Criteria:

1. Extension of disease greater than 50% of the parenchymal liver (confirmed by CAT scan or MRI)
2. Brain metastases
3. Severe and confirmed vascular diseases
4. Other concomitant malignancies except for cutaneous basal cell carcinoma or carcinoma in situ of the uterine cervix
5. Evidence of significant diseases such as uncontrolled diabetes, congestive heart failure, chronic renal insufficiency (CRI)
6. Known hypersensitivity reactions towards components of the study drugs
7. Pregnant or breastfeeding women or women of childbearing potential not making use of effective contraceptives
8. Family, psychological, social or geographical circumstances preventing the patient from undergoing follow-up and from complying with protocol procedures
9. Patients K-RAS mutant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
time to progression | one year

SECONDARY OUTCOMES:
number of adverse events | 4 months

OTHER OUTCOMES:
quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: GIAMMARIA FIORENTINI, MD, Principal Investigator — International Group of Endovascular Oncology
Locations (1):
- Azienda Ospedaliera Ospedali Riuniti Marche Nord, Presidio Ospedaliero San Salvatore, Pesaro, PU, Italy

REFERENCES:
- [Result] Fiorentini G, Aliberti C, Tilli M, Mulazzani L, Graziano F, Giordani P, Mambrini A, Montagnani F, Alessandroni P, Catalano V, Coschiera P. Intra-arterial infusion of irinotecan-loaded drug-eluting beads (DEBIRI) versus intravenous therapy (FOLFIRI) for hepatic metastases from colorectal cancer: final results of a phase III study. Anticancer Res. 2012 Apr;32(4):1387-95. PMID 22493375
- [Derived] Guadagni S, Fiorentini G, Clementi M, Palumbo P, Mambrini A, Masedu F. Mitomycin C hypoxic pelvic perfusion for unresectable recurrent rectal cancer: pharmacokinetic comparison of surgical and percutaneous techniques. Updates Surg. 2017 Sep;69(3):403-410. doi: 10.1007/s13304-017-0480-6. Epub 2017 Aug 8. PMID 28791628
- See also: International group of endovascular oncology (IGEVO) website — http://igevo.jimdo.com/